CLINICAL TRIAL: NCT04602520
Title: Dying During the Pandemic: Preserving Compassionate End-of-Life Care
Brief Title: Preserving Compassionate End of Life Care in the Pandemic
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 3WPC19
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Death; Communication, Multidisciplinary; Empathy; Compassion; Family Members; Bereavement; Empowerment; Patient Engagement
MeSH Terms: conditions — Death; Communication; Empowerment; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dying patients: Behavioral: Focused end of life conversations to promote connections among patients, family members and clinicians.
  All eligible dying patients and families in the 3 participating acute care wards are invited to participate in wish elicitation and implementation. For clinician interviews, criterion sampling will be used, based on involvement in the care of enrolled dying patients. We will use qualitative and quantitative methods to collect and analyze data. Quantitative data will include characteristics of patients, families and clinicians. Qualitative data will be based on interviews. Pending the pandemic burden, and the status of their grief, family members of deceased patients may be invited for an interview later months after the death of their loved one.
  Interventions: Behavioral: 3 Wishes Project

INTERVENTIONS:
Behavioral: 3 Wishes Project — Behavioral: Focused conversations at end-of-life to promote the connections between patients, family members, and clinicians.

SUMMARY:
Compassionate and humanistic care for patients dying in the hospital has been especially challenging during the pandemic. Family presence is restricted, maximal barrier precautions are advised, and personal protective equipment must be preserved. This research examines the impact of adaptations to compassionate approaches to end of life care in a single center.

The 3 Wishes Project (3WP) was created to promote the connections between patients, family members, and clinicians that are foundational to empathic end-of-life care. It provides a scaffold for discussions about preferences and values at the end of life and leads to acts of compassion that arise from soliciting and implementing wishes that honour the dying patient. It is partnered with the Footprints Project, which is an initiative encouraging staff to learn more about each patient. In a previous multi-center evaluation, the authors reported how the 3 Wishes Project is valuable, transferable, affordable and sustainable. During the pandemic, end of life care, facilitated by the 3 Wishes Project and Footprints Project, will be adapted to accommodate reduced family visiting and requirements to preserve PPE.

The objective of this study is to evaluate whether the adapted 3 Wishes Project continues to be feasible and valuable during the pandemic, and determine how it influences the experiences of clinicians caring for patients dying during the pandemic.

DETAILED DESCRIPTION:
This is a mixed-methods formative program evaluation of the adaptations necessitated by the pandemic to the 3 Wishes Project. The adaptations will be studied as implemented in 3 acute care units at St. Joseph's Healthcare Hamilton (medical stepdown unit, medical-surgical ICU and the COVID-19 unit) during the 2020 SARS-CoV-2 pandemic. End-of-life care for patients dying in hospital is profoundly changed during the SARS-CoV-2 pandemic, affecting the experience of everyone involved.

At this institution, end-of-life care includes 2 interventions designed to humanize the experience for patients and families (the 3 Wishes Project and Footprints Project). Both of these programs encourage clinicians to learn more about the patient as an individual and to find ways to honor them. The 3 Wishes Project is a long-running clinical program at St. Joseph's Healthcare Hamilton and has become the usual approach to end of life care, partnered with the Footprints Project which involves sharing personal information about patients with the clinical staff. In this study, to learn more about each patient, the clinical staff will telephone family members to collate personal information about patients to share with staff via a whiteboard in the patients' room, and in the patient's electronic medical record, reassuring families about interest in their loved one as a person. Building on this information about 'what matters most' and respecting and recognizing each dying patient, staff will elicit and implement terminal wishes from dying patients (if able), family members, and clinicians. During the SARS-CoV-2 pandemic, these programs will be adapted to accommodate infection prevention and control restrictions and bridge the gap when family presence is limited due to visiting restrictions.

Population: In this single-center mixed-methods formative evaluation study the researchers will enroll up to 45 patients in these 3 units, along with 45 corresponding families and 45 clinicians who cared for these patients (acknowledging that some will care for more than one dying patient). N=135 three wards in a single hospital (St. Joseph's Healthcare Hamilton)

Data: Data will be both quantitative and qualitative. Quantitative data will include patient characteristics, family visits and presence at the time of death, the number, type, and cost of terminal wishes implemented. Qualitative data will be from interviews and focus groups with clinicians and family members if not prohibited by complex grief provoked by losing a loved one during the pandemic.

ELIGIBILITY:
Inclusion Criteria (Patients):

* >18 years of age;
* >95% of dying during the hospital stay as judged by the attending physician; or
* a decision has been made to withdraw or withhold life support in anticipation of death.

Inclusion Criteria (Family Member):

- Family member or friend of dying patient

Exclusion Criteria (Patients and Family):

* Prohibitive logistical barriers (e.g., patient admitted for <24 hours);
* Patient or family declines.

N.B. A patient who has "no family" (even very broadly defined as friends and neighbours, or community members and case workers for homeless persons) would not be excluded from the wish elicitation and implementation component of the project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be admitted into the Intensive Care Unit, the Medical Step-Down unit or the Covid-19 unit who are seriously ill and have a poor outcome (>95% probability of dying during the admission). When death looms, people invariably interpret life through a lens of meaning - existential, spiritual, and relational. Through this lens, the 3 Wishes Project clearly facilitates holistic care, beyond the physical, to honor and celebrate a life. Staff are empowered and encouraged to sensitively elicit and then implementing at least 3 wishes from patients, family members, and/or clinicians caring for dying patients.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Perceptions and beliefs about value of the program | Through study completion, an average of 1 year
  Given the nascent knowledge of how the adaptations forced by the Covid-19 pandemic are perceived and experienced, it is important to understand clinician experiences of caring for dying patients during this time, and how adaptations are made to existing clinical programs designed to humanize end-of-life care. Accordingly, in this study investigators will solicit open-ended, qualitative perceptions of the value of the program. This information will be analyzed inductively to generate domains of value. Inductive analysis involves generation of categories and domains directly from the data, without pre-conceived notions of what these categories or domains might be. By generating understanding of the types of value clinicians see in this program, investigators will be able to devise ways to further refine the approach to end of life care and to measure this value in future research.
Feasibility of Enrolment as indicated by enrollment of 45 patients and successful adaptation of this approach to end of life care for all patients | Through study completion, an average of 1 year
  Enrolment will be deemed feasible when 45 patients have been enrolled and cared for with this personalized end of life care program.
Wish Implementation | Through study completion for each patient, from enrollment to 1 month postmortem
  > 3 wishes per patient are implemented; Higher proportion implemented by research and clinical staff collaboration than in pre-pandemic times.
Wish Cost of less than $5/wish | Through study completion for each patient, from enrollment to 1 month postmortem
  The $5/wish figure was established by this program in pre-pandemic times. It does not refer to patient compensation. Instead, it refers to the cost of running the intervention for each enrolled patient. Given the individually-adapted nature of this intervention, the costs will vary per participant. Affordability of the program to the unit running the program is an essential part of information collected in this program evaluation.
  Affordability will be informed by mean cost per wish and per patient at each center and overall. Also, investigators will perform a cost description of the project including both direct and indirect costs.
Family visiting as proportion of patients who had a family member present at the end of life | Through enrollment to death for each patient.
  For patients who have family or friends who desire and are able to visit, what proportion visited either physically or virtually.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Cook, MD MSc, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Participants will not be asked to consent to data sharing (qualitative or quantitative) outside the institution; further, in some instances, this would be identifying. Aggregate data will be fully reported. Feel free to contact the investigators for further information.

REFERENCES:
- [Result] Dennis B, Vanstone M, Swinton M, Brandt Vegas D, Dionne JC, Cheung A, Clarke FJ, Hoad N, Boyle A, Huynh J, Toledo F, Soth M, Neville TH, Fiest K, Cook DJ. Sacrifice and solidarity: a qualitative study of family experiences of death and bereavement in critical care settings during the pandemic. BMJ Open. 2022 Jan 19;12(1):e058768. doi: 10.1136/bmjopen-2021-058768. PMID 35046010
- [Result] Cook DJ, Takaoka A, Hoad N, Swinton M, Clarke FJ, Rudkowski JC, Heels-Ansdell D, Boyle A, Toledo F, Dennis BB, Fiest K, Vanstone M. Clinician Perspectives on Caring for Dying Patients During the Pandemic : A Mixed-Methods Study. Ann Intern Med. 2021 Apr;174(4):493-500. doi: 10.7326/M20-6943. Epub 2020 Dec 8. PMID 33284683
- [Result] Elma A, Cook D, Howard M, Takaoka A, Hoad N, Swinton M, Clarke F, Rudkowski J, Boyle A, Dennis B, Vegas DB, Vanstone M. Use of Video Technology in End-of-Life Care for Hospitalized Patients During the COVID-19 Pandemic. Am J Crit Care. 2022 May 1;31(3):240-248. doi: 10.4037/ajcc2022722. PMID 35118491